CLINICAL TRIAL: NCT00591981
Title: Preoperative Oncogeriatric Assessment for Thoracic Malignancies
Brief Title: Thoracic OncoGeriatric Assessment (TOGA) Trials
Acronym: TOGA
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: CC06504
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2015-07

CONDITIONS: Thoracic Neoplasms; Lung Neoplasms; Esophagus Neoplasms; Pleural Neoplasms; Thymus Neoplasms
Keywords: Geriatric; Thoracic; neoplasm; (Patients over 70 years of age) Geriatric oncology patients with thoracic neoplasms of the lung, esophagus, pleura and thymus.
MeSH Terms: conditions — Thoracic Neoplasms; Lung Neoplasms; Esophageal Neoplasms; Pleural Neoplasms; Thymus Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary: All patients 70 years old and above scheduled for a thoracic oncologic surgery (typically esophageal or lung cancer) will be approached for entry into this study
  Interventions: Behavioral: TOGA Tools

INTERVENTIONS:
Behavioral: TOGA Tools — ADL's, Zubrod, IADL's, BFI, MMS, MNS, GDS

SUMMARY:
Our goal is to develop a reliable, physician and patient-friendly, pre-operative Thoracic Onco-Geriatric Assessment (TOGA) to predict surgical risk in geriatric oncology patients with thoracic neoplasms of the lung, esophagus, pleura and thymus, modeled upon existing CGA tools, including the Preoperative Assessment of Cancer in the Elderly (PACE)

DETAILED DESCRIPTION:
Our proposed TOGA wil consist of portions of the PACE and some additional screening tools, and will be applied prospectively to all patients 70 years old and above seen in the UWCCC for a thoracic oncology surgery. Residents of nursing homes and assisted living facilities will be eligible for this study if they are thought to be appropriate surgical candidates; other institutionalized patients will not. The preoperative TOGA will be performed by either Drs. Weigel, Maloney, LoConte or Traynor or P.A. Block. The TOGA includes parts of the PACE, involving assessment of co-morbid illness, Activities of Daily Living [ADL], Instrumental Activities of Daily Living [IADL], Geriatric Depression Screen [GDS], Brief Fatigue Inventory [BFI], Eastern Cooperative Oncology Group/Zubrod Performance Status [PS], Mini Mental State Exam (MMSE), in addition to an American Society of Anesthesiologists Score[ASA] and mini nutritional assessment (MNA), which were not done in the PACE. The TOGA should take up to 25 minutes to complete (Audisio, 2006), and will be done at only one time preoperativelOur hypothesis is that this novel, preoperative Thoracic Onco Geriatric Assessment (TOGA) will serve to predict outcomes for older patients going though thoracic oncology surgery, and thus will enhance geriatric patient care through the development of concise, validated, preoperative risk stratification.

Our hypothesis is that this abbreviated geriatric screening tool will be a better predictor for surgical and oncologic complications after surgery than performance status alone (which is currently the only measure of fitness used in routine oncology care). In addition, we predict that parts of the TOGA, specifically the instrumental activites of daily living score (IADL), mini nutritional assessment (MNA) and the brief fatigue inventory (BFI), will be the strongest predictor(s) of outcomes in our thoracic surgery population. The outcomes data we generate will also be important in quality improvement and standardization of preoperative risk assessment for elderly patients with thoracic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients 70 years old and above seen in the UWCCC for a thoracic oncology surgery.
* Residents of nursing homes and assisted living facilities will be eligible for this study if they are thought to be appropriate surgical candidates.

Exclusion Criteria:

* Institutionalized deemed not to be appropriate.
* Prisoners

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: geriatric oncology patients with thoracic neoplasms of the lung, esophagus, pleura and thymus.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2007-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Morbidity (Cardiac, pulmonary, infectous, etc.) and Mortality in Cohort | 30days

CONTACTS AND LOCATIONS:
Overall Officials: Tracey L Weigel, MD, Principal Investigator — University of Wisconsin Dept of Surgery CardioThoracic Division
Locations (1):
- University of Wisconsin Hospital, Madison, Wisconsin, United States